CLINICAL TRIAL: NCT00723606
Title: A Randomized, Open Label, Rater Blind, Flexible Dose Multi-Center Study Comparing The Efficacy And Safety Of Intramuscular Ziprasidone With Haloperidol For Three Days In Patients With Agitation Of Schizophrenia
Brief Title: A Randomized, Open-Label, Multi-Center Study To Evaluate The Efficacy And Safety Of Intramuscular Ziprasidone In Patients With Agitation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1281152
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2010-08-25 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Schizophrenia
Keywords: Intramuscular ziprasidone, agitation, efficacy and safety
MeSH Terms: conditions — Schizophrenia; Psychomotor Agitation | interventions — ziprasidone; Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intramuscular ziprasidone (Experimental)
  Interventions: Drug: Intramuscular ziprasidone mesylate
- Intramuscular haloperidol (Active Comparator)
  Interventions: Drug: Intramuscular haloperidol

INTERVENTIONS:
Drug: Intramuscular ziprasidone mesylate — The recommended dose is 10 to 20 mg administered as required up to a maximum dose of 40 mg per day. Doses of 10 mg may be administered every two hours; doses of 20 mg may be administered every four hours up to a maximum of 40 mg/day for 3 days.
  Other Names: Zeldox, Geodon
  Arms: Intramuscular ziprasidone
Drug: Intramuscular haloperidol — The haloperidol group will receive an initial intramuscular injection of haloperidol 5mg, following on which 5mg haloperidol may be repeated every 4-8 hours to a maximum of 20 mg /day for 3 days.
  Other Names: Haldol
  Arms: Intramuscular haloperidol

SUMMARY:
This local registration study is to confirm the hypothesis of the efficacy, tolerability and safety of ziprasidone IM (intramuscular) in the Chinese population with agitation in schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese subjects aged 18-65 years (including 65) at screening.
* Subjects meeting the ICD-10 (Classification of Mental and Behavioral Disorders) criteria for schizophrenia (F20.X).
* Subjects who are in acute phase of schizophrenia and are appropriate to receive intramuscular medication for at least 3 days

Exclusion Criteria:

* History of clinically significant physical illness especially myocardial infarction, non compensatory heart failure etc.
* Subjects receiving an investigational agent in the previous 3 months prior to screening.
* Use of antipsychotic agents within 12 hours or parenteral benzodiazepines within 4 hours prior to randomization and during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- China (8):
  - Pfizer Investigational Site, Baoding, Hebei
  - Pfizer Investigational Site, Wuhan, Hubei
  - Pfizer Investigational Site, Kunming, Yunnan
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Changsha
  - Pfizer Investigational Site, Guangzhou
  - Pfizer Investigational Site, Nanjing
  - Pfizer Investigational Site, Xi'an

REFERENCES:
- [Derived] Zhang H, Wang G, Zhao J, Xie S, Xu X, Shi J, Deng H, Li K, Gao C, Wang X, Vanderburg D, Pan S, Tang H, Shu L, Karayal ON. Intramuscular ziprasidone versus haloperidol for managing agitation in Chinese patients with schizophrenia. J Clin Psychopharmacol. 2013 Apr;33(2):178-85. doi: 10.1097/JCP.0b013e3182839612. PMID 23422376
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281152&StudyName=A%20Randomized%2C%20Open-Label%2C%20Multi-Center%20Study%20To%20Evaluate%20The%20Efficacy%20And%20Safety%20Of%20Intramuscular%20Ziprasidone%20In%20Patients%20With%20Agitation

RESULTS

PARTICIPANT FLOW:
Groups:
- Ziprasidone: An initial intramuscular (IM) injection of ziprasidone 10 or 20 milligram (mg). Additional doses could have been administered according to clinical need (the total daily parenteral dose could not have exceeded 40 mg IM) for a total of 72 hours possible treatment.
- Haloperidol: An initial IM injection of haloperidol 5 mg. Following, 5 mg haloperidol could have been repeated every 4 to 8 hours to a maximum of 20 mg of haloperidol in 24 hours, depending on clinical need. The total IM treatment was continued for 72 hours.
Period: Overall Study
Arm/Group | Ziprasidone | Haloperidol
Started | 189 | 187
Completed | 185 | 180
Not Completed | 4 | 7
Not completed — Adverse Event | 2 | 5
Not completed — Other | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Ziprasidone: An initial IM injection of ziprasidone 10 or 20 mg. Additional doses could have been administered according to clinical need (the total daily parenteral dose could not have exceeded 40 mg IM) for a total of 72 hours of possible treatment.
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Haloperidol | Total
Number analyzed (Participants) | 189 | 187 | 376
Age, Customized [Number; unit: participants]
  < 18 years | 0 | 2 | 2
  18 to 44 years | 161 | 157 | 318
  45 to 64 years | 28 | 28 | 56
  > = 65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 98 | 197
  Male | 90 | 89 | 179

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Brief Psychiatric Rating Scale (BPRS) Total Scores at 72 Hours
Description: BPRS is an 18-item clinician rated scale with 11 general symptom items, 5 positive-symptom items, and 2 negative symptom items scored on a 7-point scale (1=not present and 7=extremely severe), with higher score indicating greater severity of symptom. Total possible score range=18 to 126. Change: score at final visit minus score at baseline.
Time Frame: Baseline, 72 hours
Population: Per protocol (PP) population = Full Analysis Set (FAS) subjects (ie, randomized subjects who took at least one dose of study medication) who provided a baseline and 72 hour BPRS total score and did not deviate from the protocol in a significant manner.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Haloperidol
Number analyzed (Participants) | 167 | 152
scores on a scale | -17.32 (0.692) | -18.44 (0.720)

2. Secondary Outcome: BPRS Agitation Subscale Response at 72 Hours
Description: The BPRS agitation subscale score was composed of 4 questions (questions 2, 6, 10, 17). The BPRS agitation subscale score was obtained by summing the relevant individual items. Total possible score range=4 to 28. A response was defined as a > 30 percent reduction from baseline in BPRS agitation subscale score.
Time Frame: 72 hours
Population: FAS. Missing data were replaced by last observation carried forward (LOCF).
Measure: Number; unit: participants
Arm/Group | Ziprasidone | Haloperidol
Number analyzed (Participants) | 188 | 184
participants
  Response | 149 | 155
  No Response | 39 | 29

3. Secondary Outcome: Change From Baseline in BPRS Agitation Subscale Score at 72 Hours
Description: The BPRS agitation subscale score was composed of 4 questions (questions 2, 6, 10, 17). The BPRS agitation subscale score was obtained by summing the relevant individual items. Total possible score range=4 to 28. Change: score at final visit minus score at baseline.
Time Frame: Baseline, 72 hours
Population: FAS. Missing data were replaced by LOCF.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Haloperidol
Number analyzed (Participants) | 188 | 184
scores on a scale | -6.97 (0.225) | -7.45 (0.228)

4. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score at 72 Hours
Description: CGI-I: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: 72 hours
Population: FAS. Missing data were replaced by LOCF.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Haloperidol
Number analyzed (Participants) | 188 | 184
scores on a scale | 2.52 (0.056) | 2.55 (0.057)

5. Secondary Outcome: Change From Baseline in Clinical Global Impressions Severity (CGI-S) Score at 72 Hours
Description: CGI-S: 7-point clinician rated scale to assess severity of subject's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected. Change: score at observation minus score at baseline.
Time Frame: Baseline, 72 hours
Population: FAS. Missing data were replaced by LOCF.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Haloperidol
Number analyzed (Participants) | 188 | 184
scores on a scale | -1.18 (0.061) | -1.21 (0.062)

6. Secondary Outcome: Change From Baseline in Behavioral Activity Rating Scale (BARS) at 72 Hours
Description: BARS measures the degree of agitated behavior using a 7-point scale describing increasing levels of activity (1 =difficult or unable to rouse; 2 = asleep but responds normally to verbal or physical contact; 3 = drowsy, appears sedated; 4 = quiet and awake [normal level of activity]; 5 = signs of overt [physical or verbal] activity, calms down with instructions; 6 = extremely or continuously active, not requiring restraint; 7 = violent, requires restraint.
Time Frame: Baseline, 72 hours
Population: FAS. Missing data were replaced by LOCF.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ziprasidone | Haloperidol
Number analyzed (Participants) | 186 | 185
scores on a scale | -0.93 (0.044) | -1.06 (0.044)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Ziprasidone | Haloperidol
Serious Adverse Events (participants affected / at risk) | 0/189 | 0/187
Other Adverse Events (participants affected / at risk) | 36/189 | 107/187
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=189) | Haloperidol (N=187)
Sinus tachycardia (Cardiac disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 6 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 5
Akathisia (Nervous system disorders) | 6 | 7
Dizziness (Nervous system disorders) | 7 | 6
Dystonia (Nervous system disorders) | 0 | 7
Extrapyramidal disorder (Nervous system disorders) | 4 | 69
Pyramidal tract syndrome (Nervous system disorders) | 0 | 8
Somnolence (Nervous system disorders) | 7 | 8
Insomnia (Psychiatric disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.